CLINICAL TRIAL: NCT03962647
Title: A Pilot and Feasibility Neoadjuvant Study of a 2-Week Ketogenic Diet in Combination With Letrozole to Modulate PI3K Signaling in ER+ Breast Cancer
Brief Title: A 2-Week Ketogenic Diet in Combination With Letrozole to Modulate PI3K Signaling in ER+ Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Brent Rexer, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 18108; NCI-2019-03071 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Estrogen Receptor-positive Breast Cancer
MeSH Terms: interventions — Diet, Ketogenic; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2-Week Ketogenic Diet (Experimental): 2-Week Ketogenic Diet in Combination with Letrozole
  Interventions: Dietary Supplement: 2-Week Ketogenic Diet; Drug: Letrozole
- Letrozole Control (Active Comparator)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Dietary Supplement: 2-Week Ketogenic Diet — 2-Week Ketogenic Diet in Combination with Letrozole
  Arms: 2-Week Ketogenic Diet
Drug: Letrozole — 2.5 mg taken once daily by mouth

SUMMARY:
This is a neoadjuvant study to determine the feasibility and tolerability of 2 weeks of a very low carbohydrate ketogenic diet in combination with letrozole for patients with early stage operable ER+disease.

DETAILED DESCRIPTION:
Primary Objective:

• To evaluate the feasibility and tolerability of a 2 week ketogenic diet in combination with endocrine therapy prior to surgery for early stage ER+ breast cancer.

Secondary Objectives

* To determine whether endocrine therapy in combination with a dietary intervention to reduce insulin pathway signaling results in enhanced inhibition of cancer cell proliferation (measured byKi67)
* To determine the effectiveness of 2 weeks of a ketogenic diet to reduce measures of insulin/PI3Kpathway activation in breast tumors
* To measure changes in weight and body composition after 2 weeks of a ketogenic diet
* To measure changes in insulin resistance after 2 weeks of a ketogenic diet
* To measure the effectiveness of a ketogenic diet in combination with endocrine therapy to induce and maintain a ketogenic state.

Outline:

Participants will have baseline metabolic parameters measured and will begin a 2-week diet consisting of meal replacement shakes to induce a ketogenic state. Patients will also receive letrozole 2.5 mg daily. At the end of 2 weeks, metabolic parameters will again be measured and patients will proceed with surgical treatment of their breast cancer. A tumor biopsy from the surgical specimen will be obtained to measure cell proliferation compared with the pre-treatment diagnostic biopsy.

ELIGIBILITY:
Inclusion Criteria:

* All participants must provide written informed consent.
* Patients must have histologically confirmed primary invasive mammary carcinoma

  * The tumor must be estrogen receptor positive
  * The tumor must be HER2 negative (negative IHC or FISH)
  * The primary tumor size must be at least 2 mm in size.
* Patients must be post-menopausal defined by any of the following:

  * Subjects at least 55 years of age.
  * Subjects younger than 55 years of age and amenorrheic for at least 12 months or serum follicle-stimulating hormone (FSH) levels and estradiol levels in the post-menopausal range by local lab criteria
  * Subjects with history of bilateral oophorectomy or prior radiation castration with amenorrhea for at least 6 months.
* Patients must have clinical stage I, II, or III invasive mammary carcinoma planning to undergo surgical treatment with either segmental resection or total mastectomy.
* Patients must have BMI >= 30.
* A core biopsy from the time of diagnosis must be available.
* Mammogram or ultrasound required prior to screening
* Patients must have adequate organ function based on the following laboratory parameters:

  * Serum creatinine <= 1.5x ULN
  * SGOT, SGPT <= 4x ULN (unless known steatohepatitis)
  * Serum albumin >= 2.0 g/dL
  * Total serum bilirubin <= 1.5x ULN (or <= 3x ULN if known Gilbert's syndrome)

Exclusion Criteria:

Patients with locally advanced disease who are candidates for other preoperative (chemo)therapy at the time of initial evaluation. This includes patients with inflammatory breast cancer.

* Evidence of distant metastatic disease (stage IV).
* Serious medical illness that in the judgment of the treating physician places the patient at high risk of operative mortality.
* Serious medical illness that in the judgment of the treating physician would preclude the use of a ketogenic diet.
* Severe uncontrolled malabsorption condition or disease (e.g. grade II/III diarrhea, severe malnutrition, short gut syndrome).
* Diabetes mellitus requiring insulin therapy.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Participation in any other neoadjuvant therapeutic clinical trial.
* Concurrent anti-cancer therapy other than endocrine therapy (e.g. chemotherapy, radiotherapy, immunotherapy, or any other biologic therapy).
* Concurrent treatment with an investigational agent.
* Use of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first day of dietary intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Patients who complete the dietary intervention | After 2 weeks of a ketogenic diet
  The number of patients who complete the dietary intervention, as well as the reasons for early discontinuation and any adverse events will be reported. The number of of cases where pre- and post-treatment samples could be obtained and successfully analyzed for Ki67 and insulin signaling will also be reported.

SECONDARY OUTCOMES:
Measure enhanced inhibition of cancer cell proliferation | After 2 weeks of a ketogenic diet
  Measured by Ki67
Reduction in measures of insulin/P13K pathway activation | After 2 weeks of a ketogenic diet
  Marks of insulin receptor/PI3K pathway activation in tumors
Measure changes in body composition | After 2 weeks of a ketogenic diet
  Waist circumference will be measured
Measure changes in body composition | After 2 weeks of a ketogenic diet
  Weight will be checked
Measure changes in body composition | After 2 weeks of a ketogenic diet
  Height will be checked
Measure changes in body composition | After 2 weeks of a ketogenic diet
  Body mass index will be measured
Measure changes in insulin resistance | After 2 weeks of a ketogenic diet
  Fasting glucose/insulin to measure HOMA-IR

CONTACTS AND LOCATIONS:
Overall Officials: Brent Rexer, MD, PhD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT03962647/ICF_000.pdf